CLINICAL TRIAL: NCT00961857
Title: An Open-label, Randomized Two-Part, Two-Period Crossover Study to Demonstrate the Definitive Bioequivalence After Administration of Final Market Image (FMI) Sitagliptin /Metformin 50/500 mg and 50/1000 mg Fixed Dose Combination (FDC) and Concomitant Administration of 50 mg Doses of Sitagliptin and 500 or 1000 mg Doses of Metformin as Individual Tablets
Brief Title: A Study to Demonstrate the Bioequivalence of Sitagliptin/Metformin Combination Tablets and Concomitant Administration of Sitagliptin and Metformin as Individual Tablets (0431A-048)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0431A-048; MK0431A-048; 2009_635
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Active Comparator): Individual Tablets of 50 mg sitagliptin and 500 mg metformin
  Interventions: Drug: sitagliptin phosphate (+) metformin hydrochloride; Drug: Comparator: metformin 500 mg; Drug: Comparator: sitagliptin
- Treatment B (Experimental): Sitagliptin/metformin 50 mg/500 mg tablet
  Interventions: Drug: Comparator: FMI sitagliptin/metformin 50 mg/500 mg FDC tablet
- Treatment C (Active Comparator): Individual Tablets of 50 mg sitagliptin and 1000 mg metformin
  Interventions: Drug: Comparator: sitagliptin; Drug: Comparator: metformin 1000 mg
- Treatment D (Experimental): sitagliptin/metformin 50 mg/1000 mg tablet
  Interventions: Drug: Comparator: FMI sitagliptin/metformin 50 mg/1000 mg FDC tablet

INTERVENTIONS:
Drug: sitagliptin phosphate (+) metformin hydrochloride — place holder - do not post
  Arms: Treatment A
Drug: Comparator: metformin 500 mg — A single dose of metformin 500 mg tablets
  Other Names: Apotex
  Arms: Treatment A
Drug: Comparator: sitagliptin — A single 50 mg tablet of sitagliptin
  Arms: Treatment A; Treatment C
Drug: Comparator: FMI sitagliptin/metformin 50 mg/500 mg FDC tablet — A single dose of FMI sitagliptin/metformin 50 mg/500 mg FDC tablet
  Arms: Treatment B
Drug: Comparator: FMI sitagliptin/metformin 50 mg/1000 mg FDC tablet — A single dose of FMI sitagliptin/metformin 50 mg/1000 mg FDC tablet
  Arms: Treatment D
Drug: Comparator: metformin 1000 mg — A single dose of metformin 1000 mg tablets
  Other Names: Apotex
  Arms: Treatment C

SUMMARY:
A two-part study to demonstrate the bioequivalence of a single dose of the Final Market Image (FMI) of sitagliptin /metformin (50/500 and 50/1000 mg) Fixed-Dose Combination (FDC) tablet and co-administration of a single dose of sitagliptin (50 mg) and metformin ( 500 or 1000 mg) as individual tablets. Subject will only participate in one part, receiving treatment A and B (Part I) or Treatment C and D (Part II).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of reproductive potential test negative for pregnancy and agree to use appropriate contraception
* Subject is in good health and is a non-smoker
* Subject is willing to avoid strenuous physical activity during the study
* Subject agrees to refrain from eating grapefruit or grapefruit products during the study

Exclusion Criteria:

* Subject has a history of neoplastic disease (cancer), stroke, chronic seizures, or major neurological disorder. Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Subject consumes excessive amounts of alcohol or caffeinated beverages
* Subject has donated blood, had surgery or participated in another clinical study within the past 4 weeks
* Subject has a history of significant multiple and/or severe allergies to prescription or non-prescription drugs or food
* Subject has a history of hypersensitivity to metformin, sitagliptin, or sitagliptin/Metformin
* Subject is a regular user or past abuser of any illicit drugs
* Subject is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies during the study.
* Subject is a nursing mother

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2005-12-01 (Actual); Study Completion 2006-01-01 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration vs. time curve (AUC) after administration of sitagliptin/metformin (50/500 and 50/1000 mg/mg) FDC tablet and co-administration of corresponding doses of sitagliptin and metformin as individual tablets | 72 hours post dose

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of sitagliptin and metformin after administration of sitagliptin/metformin (50/500 and 50/1000 mg/mg) FDC tablet and co-administration of corresponding doses of sitagliptin and metformin as individual tablets | 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Migoya EM, Miller JL, Gutierrez M, Zheng W, Johnson-Levonas AO, Liu Q, Matthews CZ, Wagner JA, Gottesdiener KM. Bioequivalence of sitagliptin/metformin fixed-dose combination tablets and concomitant administration of sitagliptin and metformin in healthy adult subjects: a randomized, open-label, crossover study. Clin Drug Investig. 2010;30(12):855-66. doi: 10.1007/BF03256914. PMID 20923244